## **COVER PAGE**

Official Title of the Study: Maternal Cognitive Function and Neurobehavioral

**Development of Underprivileged Children** 

NCT Number : NCT03321591

Date of the Document : 19/09/2016

**Statistical Analysis Plan**: Data will be analyzed by using correlation and multiple regression analysis in order to see the relationship between maternal cognitive function and neurobehavioral development of children. Furthermore, I have a plan to use path analysis (structural equation modeling). In this regard, I have prepared a model to test as under. It is very tough and time consuming to test model fit equation. I have to study more and more on the books of statistics and experts to handle LISREL or SPSS AMOS software.

